CLINICAL TRIAL: NCT01925274
Title: A RANDOMIZED PHASE 2 STUDY OF PF-05212384 PLUS IRINOTECAN VERSUS CETUXIMAB PLUS IRINOTECAN IN PATIENTS WITH KRAS AND NRAS WILD TYPE METASTATIC COLORECTAL CANCER
Brief Title: A Study Of PF-05212384 Plus Irinotecan Vs Cetuximab Plus Irinotecan In Patients With KRAS And NRAS Wild Type Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment to the study was terminated on 11Nvo2014 due to slow recruitment. There were no safety or efficacy issues that contributed to this decision.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2151005; 2013-002095-40 (EudraCT Number)
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; colorectal cancer; KRAS; colon cancer; mCRC; CRC; PF-05212384; KRAS wild type colorectal cancer; irinotecan; cetuximab; NRAS
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — gedatolisib; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): PF-05212384 plus Irinotecan
  Interventions: Drug: PF-05212384; Drug: irinotecan
- Arm B (Active Comparator): Cetuximab plus Irinotecan
  Interventions: Drug: Cetuximab; Drug: Irinotecan

INTERVENTIONS:
Drug: PF-05212384 — 30 minute IV infusion of PF-05212384 on days 2, 9, 16 and 23 of each cycle. Intra-patient dose escalation will commence with 110mg and will increase depending on tolerability.
  Other Names: PKI-587
  Arms: Arm A
Drug: irinotecan — 90 minutes IV infusion of irinotecan 180mg/m^2 on days 1 and 15 of each cycle
  Other Names: Camptosar, Campto, CPT-11
  Arms: Arm A
Drug: Cetuximab — 120 minute IV infusion of cetuximab 400mg/m^2 on cycle 1 day 1; 60 minute IV infusion of cetuximab on days 8, 15, and 22 of each cycle, and on day 1 of each cycle after cycle 1
  Other Names: Erbitux
  Arms: Arm B
Drug: Irinotecan — 90 minutes IV infusion of Irinotecan 180mg/m^2 on days 1 and 15 of each cycle
  Other Names: Camptosar, Campto, CPT-11
  Arms: Arm B

SUMMARY:
This study will investigate whether the combination of PF-05212384 plus Irinotecan improves progression free survival in patients with KRAS and NRAS wild type metastatic colorectal cancer when compared with the combination of cetuximab plus Irinotecan. A Japanese Lead in Cohort will assess the safety of the combination of PF-05212384 + irinotecan in patients enrolled at Japanese sites.

ELIGIBILITY:
Inclusion Criteria:

* KRAS and NRAS wild type metastatic colorectal cancer
* Progression following treatment for colorectal cancer with irinotecan, oxaliplatin and fluoropyrimidine therapy in the metastatic setting.
* Eastern Cooperative Oncology Group [ECOG] Performance Status of 0, 1, or 2
* At least one measurable lesion by Response Evaluation Criterion in Solid Tumors [RECIST]

Exclusion Criteria:

* More than 2 prior cytotoxic chemotherapy regimens for metastatic colorectal cancer.
* Prior treatment with a PI3K, mTOR, AKT or EGFR inhibitor
* Patients who have discontinued treatment with prior irinotecan therapy due to toxicity.
* Prior radiation to the pelvis or abdomen
* Patients with history of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (22):
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Drug Management Only: UCLA West Medical Pharmacy, Att: Steven L Wong, Pharm D, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Los Angeles, California
  - UCLA West Medical Pharmacy, Los Angeles, California
  - Regulatory Management Only: TRIO-US Central Administration, Los Angeles, California
  - TRIO-US Central Administration (Regulatory Management only), Los Angeles, California
  - TRIO_US, Los Angeles, California
  - West Valley Hematology/Oncology Med Group, Northridge, California
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Regulatory Office: Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Kadlec Medical Center, Richland, Washington
  - Outpatient Imaging Center, Richland, Washington
  - Medical Oncology Associates, PS, Spokane, Washington
  - Spokane Valley Cancer Center, Spokane Valley, Washington
- Japan (2):
  - Aichi cancer center central hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
- South Korea (4):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital / Department of Internal Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2151005&StudyName=A%20Study%20Of%20PF-05212384%20Plus%20Irinotecan%20Vs%20Cetuximab%20Plus%20Irinotecan%20In%20Patients%20With%20KRAS%20And%20NRAS%20Wild%20Type%20Metastatic%20Colorectal%20Can

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-05212384 + Irinotecan: Arm A: PF-05212384 was administered intravenously (IV) every week (Days 2, 9, 16 and 23 of each 28-day cycle) at a starting dose level of 110 mg. During Cycle 1, PF-05212384 was only dosed on Days 9, 16 and 23. After one cycle of dosing with PF-05212384, in subsequent cycles, the dose level remained at 110 mg or was escalated based on the occurrences of dose limiting toxicities (DLTs) in previous cycle and at the discretion of the investigator. Participants enrolled in Korea remained at the 110 mg starting dose level of PF-05212384. Irinotecan was administered IV every other week (Days 1 and 15 of each 28-day cycle) at a dose level of 180 mg/m^2. Both the dose levels of PF-05212384 and irinotecan were adjusted according to severity of toxicities. Infusion of PF-05212384 followed irinotecan infusion by at least 24 hours (+/- 10%).
- Cetuximab + Irinotecan: Arm B: Cetuximab was administered IV every week (Days 1, 8, 15 and 22 of each 28-day cycle) at a starting dose level of 400 mg/m^2 on Cycle 1 Day 1 followed by 250 mg/m^2 in subsequent infusions. Irinotecan was administered IV every other week (Days 1 and 15 of each 28-day cycle) at a dose level of 180 mg/m^2. Both the dose levels of cetuximab and irinotecan were adjusted according to severity of toxicities.
- PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC): PF-05212384 was administered intravenously (IV) every week (Days 2, 9, 16 and 23 of each 28-day cycle) at a starting dose level of 110 mg. During Cycle 1, PF-05212384 was only dosed on Days 9, 16 and 23. Irinotecan was administered IV every other week (Days 1 and 15 of each 28-day cycle) at a dose level of 180 mg/m^2. Both the dose levels of PF-05212384 and irinotecan were adjusted according to severity of toxicities. Infusion of PF-05212384 followed irinotecan infusion by at least 24 hours (+/- 10%).
Period: Overall Study
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Started | 7 | 6 | 6
Completed | 0 | 0 | 0
Not Completed | 7 | 6 | 6
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Study terminated by sponsor | 4 | 0 | 0
Not completed — Protocol amendment | 1 | 3 | 6

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all enrolled participants who received the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC) | Total
Number analyzed (Participants) | 7 | 6 | 6 | 19
Age, Customized [Number; unit: participants]
  <18 years | 0 (7.8) | 0 (6.1) | 0 (6.7) | 0
  18-64 years | 5 | 4 | 4 | 13
  >=65 years | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 11
  Male | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Investigators
Description: Progression-free survival (PFS) was the time from the first dose of study treatment to the first documentation of objective tumor progression or death due to any cause, whichever occurred first. Objective progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. Median PFS was estimated based on the Kaplan-Meier method.
Time Frame: From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
Population: All participants who were randomized, with KRAS (Kirsten ras oncogene) and NRAS (neuroblastoma ras viral oncogene homolog) wild type status confirmed by central lab, and with treatment arm assignment designated according to randomization. As pre-specified in the protocol, this outcome measure was not analyzed for Japanese Lead-In Cohort.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B
Number analyzed (Participants) | 4 | 3
months | 3.7 [1.5 to 7.4] | NA [NA to NA] — Less than 50% of the population experienced an event, therefore, median and 95% confidence interval were not calculated. The only individual value was 16.6 months.

2. Secondary Outcome: Number of Participants With Unacceptable Toxicity in Cycle 1 (Japanese LIC Only)
Description: Unacceptable toxicity (according to Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0) was any of the following occurrences: (1) Grade 4 neutropenia >7 days, or febrile neutropenia, or Grade 4 thrombocytopenia; (2) Grade >=3 nausea/vomiting despite optimal antiemetic treatment, or Grade >=3 diarrhea despite optimal anti diarrheal treatment; (3) unmanageable Grade >=3 hyperglycemia; (4) mean QTc interval (time from electrocardiogram [ECG] Q wave to the end of the T wave corresponding to electrical systole, corrected for heart rate) >501 msec in triplicate 12-lead ECG, or myocardial infarction, or ventricular arrhythmia; (5) Grade >=3 non-hematologic toxicity; (6) treatment delay of >=2 weeks due to study drug related toxicity; (7) persistent, intolerable toxicities which resulted in failure to deliver at least 75% of doses of both PF-05212384 and irinotecan during Cycle 1; (8) Grade >=2 respiratory toxicities.
Time Frame: 28 days
Population: The analysis population included all participants enrolled into Japanese LIC. As pre-specified in protocol, this outcome measure was not analyzed for reporting arms: "PF-05212384 + Irinotecan: Arm A" and "Cetuximab + Irinotecan: Arm B".
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6
participants | 0

3. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response was based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1. Confirmed PR was defined as disappearance of all target lesions. Confirmed PR was defined as >=30% decrease in sum of the longest dimensions of the target lesions taking the baseline sum as a reference. Confirmed responses were those that persisted on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: 2 years
Population: Response evaluable analysis set was used for the analysis of objective response, and it included all participants in the full analysis set (all participants who were randomized, with treatment arm assignment designated according to randomization) who had an adequate baseline assessment of disease and measurable disease.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
percentage of participants | 14.3 [0.4 to 57.9] | 50.0 [11.8 to 88.2] | 0 [0.0 to 45.9]
Statistical Analysis 1: Comparison: PF-05212384 + Irinotecan: Arm A vs Cetuximab + Irinotecan: Arm B; Test type: Superiority or Other; p = 0.164, Chi-squared; Mean Difference (Net) = -35.71, 95% CI 2-sided [-83.4 to 12.0]

4. Secondary Outcome: Duration of Response
Description: For participants with an objective response (CR or PR), duration of response was defined as the time from first documentation of CR or PR to date of first documentation of objective progression or death. Date of first documentation of progression and date of first documentation of CR or PR were based on Investigator's assessment of response.
Time Frame: 2 years
Population: The analysis population included all participants who achieved CR or PR in Arm A and Arm B. As pre-specified in protocol, this outcome measure was not analyzed for reporting arm "PF 05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)".
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B
Number analyzed (Participants) | 1 | 3
months | NA [NA to NA] — Only 1 participant achieved CR or PR, therefore, median and 95% confidence interval were not calculated. The only individual value was 5.6 months. | NA [NA to NA] — Less than 50% of the population experienced subsequent progression or death, therefore, median and 95% confidence interval were not calculated. The only individual value was 14.8 months.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the duration from enrollment to death. Participants last known to be alive were censored at date of last contact.
Time Frame: 2 years
Population: Per protocol analysis set, i.e. all participants who were randomized, with KRAS and NRAS wild type status confirmed by central lab and with treatment arm assignment designated according to randomization. As pre-specified in protocol, this outcome measure was not analyzed for reporting arm "PF 05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)".
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B
Number analyzed (Participants) | 4 | 3
months | NA [3.3 to NA] — Median was not calculated, since less than 50% of population died. | NA [NA to NA] — No death occurred in this arm.

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE was defined as any untoward occurrence at any dose that resulted in death; was life threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect. AEs included both serious and non-serious AEs. Treatment-emergent AEs were those with initial onset or increasing in severity after the first dose of study drug.
Time Frame: Administration of the first dose of study drug through 28 calendar days after the last administration of study drug
Population: Safety analysis set included all participants who received at least one dose of study treatment, with treatment arm assignment designated according to actual study treatment received.
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  AEs | 7 | 6 | 6
  SAEs | 3 | 1 | 1

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: TEAEs were those AEs with initial onset or increasing in severity after the first dose of study drug. CTCAE version 4.0 was used to grade the severity of TEAEs. Grade 1 referred to mild AEs; Grade 2 referred to moderate AEs; Grade 3 referred to severe AEs; Grade 4 referred to AEs with life-threatening consequences, and urgent intervention was needed to manage them; Grade 5 referred to death related to AE.
Time Frame: Administration of the first dose of study drug through 28 calendar days after the last administration of study drug
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  Grade 1 | 1 | 2 | 2
  Grade 2 | 1 | 1 | 0
  Grade 3 | 3 | 2 | 4
  Grade 4 | 2 | 0 | 0
  Grade 5 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Laboratory Test (Hematology) Abnormalities
Description: The following hematology parameters were evaluated in this study: hemoglobin, white blood cells (WBC) with differential, and platelets.
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  Anemia | 6 | 6 | 6
  Hemoglobin increased | 0 | 0 | 0
  Lymphocyte count increased | 0 | 2 | 0
  Lymphopenia | 5 | 4 | 5
  Neutrophils (absolute) | 4 | 3 | 5
  Platelets | 0 | 3 | 1
  White blood cells | 4 | 4 | 5

9. Secondary Outcome: Number of Participants With Laboratory Test (Chemistry) Abnormalities
Description: The following chemistry parameters were evaluated in this study: sodium, potassium, magnesium, chloride, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin, albumin, blood urea nitrogen (BUN) or urea, creatinine, total calcium, glycosylated hemoglobin (HbA1c), glucose, uric acid, phosphorus or phosphate, insulin, and C-peptide.
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  ALT | 2 | 1 | 1
  Alkaline phosphatase | 3 | 4 | 4
  AST | 2 | 1 | 1
  Total bilirubin | 0 | 1 | 0
  Creatitine | 4 | 3 | 6
  Hypercalcemia | 1 | 0 | 0
  Hyperglycemia | 6 | 4 | 4
  Hyperkalemia | 1 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0
  Hypernatremia | 1 | 0 | 1
  Hypoalbuminemia | 2 | 4 | 4
  Hypocalcemia | 2 | 3 | 3
  Hypoglycemia | 0 | 1 | 0
  Hypokalemia | 2 | 2 | 3
  Hypomagnesemia | 3 | 4 | 1
  Hyponatremia | 2 | 1 | 0
  Hypophosphatemia | 2 | 1 | 0

10. Secondary Outcome: Number of Participants With Laboratory Test (Urinalysis) Abnormalities
Description: Urinalysis included urine dipstick for protein and blood: if positive, perform a microscopic analysis. Number of participants with urine protein tested positive is presented.
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants | 3 | 1 | 4

11. Secondary Outcome: Number of Participants With Laboratory Test (Coagulation) Abnormalities
Description: Coagulation analysis included partial thromboplastin time (PTT) and international normalized ratio (INR) or prothrombin time (PT).
Time Frame: 2 years
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  PTT (number of participants =7, 6, 5) | 2 | 4 | 0
  PT (number of participants =7, 5, 6) | 3 | 3 | 1
  PT INR | 1 | 2 | 2

12. Secondary Outcome: Number of Participants With ECG Post-Baseline Maximum Absolute Values Meeting Pre-defined Criteria
Description: The number of participants with ECG post-baseline maximum absolute values meeting the following criteria was reported: (1) maximum QTc interval ranged from 450 to 480 msec; >480-500 msec; >500 msec; (2) maximum QTcB (QT corrected for heart rate using Bazett's formula) interval ranged from 450 to 480 msec; >480-500 msec; >500 msec; (3) maximum QTcF (QT corrected for heart rate using Fridericia's formula) interval ranged from 450 to 480 msec; >480-500 msec; >500 msec.
Time Frame: 2 years
Population: QTc analysis set included all participants in the safety analysis set who had at least one ECG assessment after receiving study treatment.
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 3 | 6
participants
  Maximum QTc interval: 450-480 msec | 2 | 1 | 1
  Maximum QTc interval: >480-500 msec | 0 | 0 | 0
  Maximum QTc interval: >500 msec | 0 | 0 | 0
  Maximum QTcB interval: 450-480 msec | 3 | 1 | 0
  Maximum QTcB interval: >480-500 msec | 0 | 0 | 0
  Maximum QTcB interval: >500 msec | 0 | 0 | 0
  Maximum QTcF interval: >450-480 msec | 1 | 0 | 0
  Maximum QTcF interval: >480-500 msec | 0 | 0 | 0
  Maximum QTcF interval: >500 msec | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With ECG Maximum Increase From Baseline Meeting Pre-defined Criteria
Description: The number of participants with ECG maximum increase from baseline meeting the following criteria was reported:
  Criterion A: maximum QTc interval increase from baseline >30 msec and ≤60 msec; criterion B: maximum QTc interval increase from baseline >60 msec; criterion C: maximum QTcB interval increase from baseline >30 msec and ≤60 msec; criterion D: maximum QTcB interval increase from baseline >60 msec; criterion E: maximum QTcF interval increase from baseline >30 msec and ≤60 msec; criterion F: maximum QTcF interval increase from baseline >60 msec.
Time Frame: 2 years
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 3 | 6
participants
  Criterion A | 1 | 1 | 0
  Criterion B | 0 | 0 | 0
  Criterion C | 0 | 1 | 0
  Criterion D | 0 | 0 | 0
  Criterion E | 0 | 0 | 0
  Criterion F | 0 | 0 | 0

14. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-05212384
Description: Cmax of PF-05212384 was observed directly from data.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 24, 72, 120 hours post PF-05212384 infusion on Cycle 1 Day 9 and Cycle 1 Day 16.
Population: The pharmacokinetic concentration analysis set included all randomized participants (or enrolled participants to the Japanese LIC) who started treatment and had at least one time point with a concentration measurement recorded. As pre-specified in protocol, this outcome measure was not analyzed for reporting arm: "Cetuximab + Irinotecan: Arm B".
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 6
ng/mL
  Cycle 1 Day 9 | 8345 (19) | 8534 (10)
  Cycle 1 Day 16 (number of participants =5, 6) | 10120 (27) | 9670 (26)

15. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Irinotecan
Description: Cmax of irinotecan was observed directly from data.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
ng/mL
  Cycle 1 Day 1 | 2283 (30) | 2123 (18)
  Cycle 2 Day 1 (number of participants =4, 5) | 1620 (41) | 1999 (13)

16. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SN-38
Description: SN-38 is an irinotecan metabolite. Cmax of SN-38 was observed directly from data.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
ng/mL
  Cycle 1 Day 1 | 23.51 (32) | 24.25 (50)
  Cycle 2 Day 1 (number of participants =4, 5) | 22.81 (67) | 28.04 (33)

17. Secondary Outcome: Time for Maximum Plasma Concentration (Tmax) of PF-05212384
Description: Tmax of PF-05212384 was observed directly from data as time of first occurrence.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 24, 72, 120 hours post PF-05212384 infusion on Cycle 1 Day 9 and Cycle 1 Day 16.
Population: The pharmacokinetic parameter analysis set included all randomized participants (or enrolled participants to the Japanese LIC) who started treatment and had at least one of the pharmacokinetic parameters of interest estimated. As pre-specified in protocol, this outcome measure was not analyzed for reporting arm: "Cetuximab + Irinotecan: Arm B".
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 6
hours
  Cycle 1 Day 9 | 0.483 [0.467 to 0.517] | 0.483 [0.467 to 0.500]
  Cycle 1 Day 16 (number of participants =5, 6) | 0.500 [0.467 to 0.517] | 0.500 [0.483 to 0.517]

18. Secondary Outcome: Time for Maximum Plasma Concentration (Tmax) of Irinotecan
Description: Tmax of irinotecan was observed directly from data as time of first occurrence.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
hours
  Cycle 1 Day 1 | 1.50 [1.47 to 1.62] | 1.53 [1.48 to 1.58]
  Cycle 2 Day 1 (number of participants =4, 5) | 1.55 [1.50 to 2.05] | 1.53 [1.50 to 1.57]

19. Secondary Outcome: Time for Maximum Plasma Concentration (Tmax) of SN-38
Description: SN-38 is an irinotecan metabolite. Tmax of SN-38 was observed directly from data as time of first occurrence.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: The pharmacokinetic parameter analysis set included all randomized participants (or enrolled participants to the Japanese LIC) who started treatment and had at least one of the pharmacokinetic parameters of interest estimated. As pre specified in protocol, this outcome measure was not analyzed for reporting arm: "Cetuximab + Irinotecan: Arm B".
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
hours
  Cycle 1 Day 1 | 2.00 [1.50 to 2.18] | 1.98 [1.48 to 2.08]
  Cycle 2 Day 1 (number of participants =4, 5) | 2.03 [1.53 to 3.98] | 1.93 [1.90 to 2.00]

20. Secondary Outcome: Terminal Elimination Half Life (t½) of PF-05212384
Description: T½ was calculated as loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 24, 72, 120 hours post PF-05212384 infusion on Cycle 1 Day 9 and Cycle 1 Day 16.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 6
hours
  Cycle 1 Day 9 | 37.65 (4.55) | 37.78 (3.61)
  Cycle 1 Day 16 (number of participants =4, 6) | 35.10 (6.90) | 36.07 (4.56)

21. Secondary Outcome: Terminal Elimination Half Life (t½) of Irinotecan
Description: as for outcome 20
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
hours
  Cycle 1 Day 1 | 5.547 (0.562) | 5.255 (0.420)
  Cycle 2 Day 1 (number of participants =4, 5) | 5.293 (0.488) | 5.344 (0.719)

22. Secondary Outcome: Terminal Elimination Half Life (t½) of SN-38
Description: as for outcome 20
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 2 | 4
hours
  Cycle 1 Day 1 (number of participants =2, 3) | NA (NA) — These summary statistics were not calculated, as the number of participants being analyzed was fewer than 3, considered as non-reliable for analysis. The individual values of these two participants were 8.05 and 8.56 hours, respectively. | 9.890 (0.811)
  Cycle 2 Day 1 | NA (NA) — These summary statistics were not calculated, as the number of participants being analyzed was fewer than 3, considered as non-reliable for analysis. The individual values of these two participants were 8.44 and 8.74 hours, respectively. | 8.840 (1.091)

23. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero to the Time for the Last Quantifiable Concentration (AUClast) of PF-05212384
Description: AUClast refers to the area under plasma concentration time profile from time zero to the time for the last quantifiable concentration. AUClast of PF-05212384 was determined using linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 24, 72, 120 hours post PF-05212384 infusion on Cycle 1 Day 9.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 11530 (15) | 13390 (17)

24. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero to the Time for the Last Quantifiable Concentration (AUClast) of Irinotecan
Description: AUClast refers to the area under plasma concentration time profile from time zero to the time for the last quantifiable concentration. AUClast of irinotecan was determined using linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
ng*hr/mL
  Cycle 1 Day 1 | 11860 (23) | 11030 (29)
  Cycle 2 Day 1 (number of participants =4, 5) | 8776 (62) | 10380 (29)

25. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero to the Time for the Last Quantifiable Concentration (AUClast) of SN-38
Description: AUClast refers to the area under plasma concentration time profile from time zero to the time for the last quantifiable concentration. AUClast of SN-38 (an irinotecan metabolite) was determined using linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
ng*hr/mL
  Cycle 1 Day 1 | 217.0 (29) | 217.9 (38)
  Cycle 2 Day 1 (number of participants =4, 5) | 182.4 (43) | 228.5 (38)

26. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-05212384
Description: AUCinf refers to the area under plasma concentration time profile from time zero extrapolated to infinite time. AUCinf of PF-05212384 was calculated using the formula: AUCinf = AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 24, 72, 120 hours post PF-05212384 infusion on Cycle 1 Day 9.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 11700 (15) | 13580 (17)

27. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Irinotecan
Description: AUCinf refers to the area under plasma concentration time profile from time zero extrapolated to infinite time. AUCinf of irinotecan was calculated using the formula: AUCinf = AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6
ng*hr/mL
  Cycle 1 Day 1 | 12480 (23) | 11570 (30)
  Cycle 2 Day 1 (number of participants =4, 5) | 9216 (63) | 10950 (31)

28. Secondary Outcome: Area Under Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of SN-38
Description: AUCinf refers to the area under plasma concentration time profile from time zero extrapolated to infinite time. AUCinf of SN-38 (an irinotecan metabolite) was calculated using the formula: AUCinf = AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: Pre-dose (0 hour), 1.5, 2, 4, 6 and 24 hours post irinotecan infusion on Cycle 1 Day 1 and Cycle 2 Day 1.
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-05212384 + Irinotecan: Arm A | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 2 | 4
ng*hr/mL
  Cycle 1 Day 1 (number of participants =2, 3) | NA (NA) — These summary statistics were not calculated, as the number of participants being analyzed was fewer than 3, considered as non-reliable for analysis. The individual values of these two participants were 218 and 218 ng*hr/mL, respectively. | 230.4 (13)
  Cycle 2 Day 1 | NA (NA) — These summary statistics were not calculated, as the number of participants being analyzed was fewer than 3, considered as non-reliable for analysis. The individual values of these two participants were 120 and 215 ng*hr/mL, respectively. | 279.7 (45)

29. Secondary Outcome: Levels of Signaling Proteins in Paired and Single Tumor Biopsies
Description: Pre defined signaling proteins included Akt (protein kinase B), p-Akt (phosphorylated Akt), p-S6 (phosphorylated ribosomal protein S6), p-Met (phosphorylated Met, a receptor tyrosine kinase), p-mTOR (phosphorylated mammalian target of rapamycin), EGFR (epithelial growth factor receptor), and p-EGFR (phosphorylated EGFR).
Time Frame: 2 years
Population: Data for this outcome measure were not collected due to early termination of this study.
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Expression of Pre-defined Gene Sequences in Biopsied Tumor Tissues
Description: Pre-defined gene sequences were those related to EGFR, PI3K (phosphoinositide-3 kinase) and other oncogenic pathways; examples included but were not limited to PIK3CA (this gene encodes the catalytic subunit of PI3K), PIK3R1 (this gene encodes the regulatory subunit of PI3K), KRAS, NRAS and BRAF (this gene encodes serine/threonine-protein kinase B-Raf) sequences and PIK3CA gene amplification. Due to early termination of this study, these pre-defined gene sequences were not analyzed, except for KRAS and NRAS. Number of participants who had KRAS and NRAS wild type status confirmed by the central laboratory is presented.
Time Frame: 2 years
Population: All participants for whom at least one of these pre-defined gene sequences was analyzed were included.
Measure: Number; unit: participants
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Number analyzed (Participants) | 7 | 6 | 6
participants
  Confirmed wild type KRAS | 4 | 3 | 6
  Confirmed wild type NRAS | 4 | 3 | 3

31. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Colorectal (FACT-C)
Description: Functional Assessment of Cancer Therapy-Colorectal (FACT-C) was used in this study to assess Health-Related Quality of Life (HRQoL) and CRC-related symptoms in participants enrolled to the randomized portion of the study. The FACT-C is part of the Functional Assessment of Chronic Illness Therapy (FACIT) measurement system, a comprehensive and extensive set of self-reported instruments for the assessment of health-related quality of life in participants with cancer or other chronic illnesses.
Time Frame: 2 years
Population: Data for this outcome measure were no longer collected after approval of protocol amendment 4, and data previously collected were insufficient to perform any analysis.
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC): PF-05212384 was administered intravenously (IV) every week (Days 2, 9, 16 and 23 of each 28-day cycle) at a starting dose level of 110 mg. During Cycle 1, PF-05212384 was only dosed on Days 9, 16 and 23. Irinotecan was administered IV every other week (Days 1 and 15 of each 28 day cycle) at a dose level of 180 mg/m^2. Both the dose levels of PF 05212384 and irinotecan were adjusted according to severity of toxicities. Infusion of PF-05212384 followed irinotecan infusion by at least 24 hours (+/- 10%).
Arm/Group | PF-05212384 + Irinotecan: Arm A | Cetuximab + Irinotecan: Arm B | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC)
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/6 | 1/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05212384 + Irinotecan: Arm A (N=7) | Cetuximab + Irinotecan: Arm B (N=6) | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC) (N=6)
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-05212384 + Irinotecan: Arm A (N=7) | Cetuximab + Irinotecan: Arm B (N=6) | PF-05212384 + Irinotecan: Japanese Lead-In Cohort (LIC) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 3
Stomatitis (Gastrointestinal disorders) | 5 | 1 | 4
Vomiting (Gastrointestinal disorders) | 4 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 1
Influenza like illness (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 2
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated by sponsor due to strategic reasons and not due to any safety or efficacy concerns with treatment of PF-05212384.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.